CLINICAL TRIAL: NCT02163720
Title: Non Interventional Study Dealing With the Use of Trabectedin (Yondelis®)-Pegylated Liposomal Doxorubicin (Caelyx®) in Patient With Platinum-sensitive Relapse
Brief Title: Ovarian Cancer Treatment Platinum-sensitive Relapse - Cohort Study (PROSPECTYON)
Status: Completed | Type: Observational
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Other Study IDs: PROSPECTYON (GINECO-OV229)
Record Dates: First submitted 2014-05-28; First posted 2014-06-16 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; fallopian tube or primary peritoneal; relapse; platinum-sensitive; Yondelis®-Caelyx®
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Yondelis®-Caelyx®-relapse ovarian cancer: Yondelis®-Caelyx®-relapse ovarian cancer
  Interventions: Drug: Yondelis®-Caelyx®

INTERVENTIONS:
Drug: Yondelis®-Caelyx® — Observation of Yondelis®-Caelyx® administration
  Other Names: Observation of Yondelis®-Caelyx® administration

SUMMARY:
The French cooperative group GINECO proposes to implement an observational study to describe a real situation, in daily practice tolerance and methods of administration of trabectedin (Yondelis®)-Pegylated liposomal doxorubicin(Caelyx)®, in ovarian platinum sensitive cancer relapse.

DETAILED DESCRIPTION:
Population : Patients aged 18 years and older with an epithelial ovarian cancer, fallopian tube or primary peritoneal with platinum-sensitive recurrent witch it was decided to initiate a treatment with trabectedin (Yondelis®)-Pegylated liposomal doxorubicin(Caelyx)®.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over,
* Patients with an epithelial ovarian cancer, fallopian tube or peritoneal who will receive Yondelis®-Caelyx® in relapse platinum-sensitive
* Patients should be informed of the study orally and should not have any objection their data to be processed

Exclusion Criteria:

* Patient participation in a clinical trial
* Patient non-affiliated to a social security scheme.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with epithelial ovarian cancer, fallopian tube or peritoneal with treatment receiving in relapse platinum-sensitive
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2014-07-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
Evaluate the proportion of patient partially versus fully platinum-sensitive in relapse ovarian cancer | Patient will be followed during 12 months
  To assess patient safety and the tolerance of Yondelis®-Caelyx® administered regarding the daily practice of the oncologist.

SECONDARY OUTCOMES:
Choice of treatment | at baseline
  Describe the reason why treatment by trabectedin and doxorubicine combination was initiated (ex : number of patients with previous intolerance to platinum as allergic reaction, residual peripherical neuropathy, alopecia; availability of the combination yondelis-caelyx in the treating site; number of sites where the yondelis-caelyx combination is the reference treatment)
Characteristics of the population registered | at baseline
  Describe the population that will be registered
Evaluation of the modality of use of Yondelis®-Caelyx® | during treatment (expected period = 6 months)-As it is an non interventionnal study, treatment period corresponds to the routine practice of each investigator
  Describe the way how treatment by Yondelis®-Caelyx® is administered in the daily practice for each patient (Initial dosage of caelyx and yondelis, number of cycles administered for each treatment , dose reductions occurence and reasons)
Safety according to CTCAE v4.03 criteria | Patient will be followed during 12 months
  To assess patient safety and the tolerance of Yondelis®-Caelyx® administered regarding the daily practice of the oncologist.
Evaluation of clinical benefit | baseline and during treatment (expected period of treatment = 6 months). As it is an non interventionnal study, treatment period corresponds to the routine practice of each investigator.
  Evaluation of clinical benefit will be performed during the physical examination at baseline and during the treatment
  At baseline : describe the number of patients how present the following related symptom disease : weight loss, ascites, abdominal pain, constipation, fatigue, occlusive syndrome
  Then, describe the number of patients how presented and improvement or a degradation of theses related symptom disease during the treatment
  Nota Bene : this cohort study is strictly observational and must represent the daily practice. No indications must be given regarding the frequency of the physical examination
Efficacy of treatments | during treatment and follow up period (maximum of 12 months)
  Evaluate the efficacy of Yondelis®-Caelyx® in terms of progression-free survival (PFS), Overall Survival (OS), response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric SELLE, MD, Principal Investigator — Hôpital Tenon
Locations (33):
- France (33):
  - Centre de Radiothérapie et d'Oncologie, Agen
  - Clinique de l'Europe, Amiens
  - ICO Paul Papin, Angers
  - Hôpital de la Côte Basque, Bayonne
  - Hôpital jean Minjoz, Besançon
  - Clinique Tivoli, Bordeaux
  - Hôpital Fleyriat, Bourg-en-Bresse
  - Hôpital Morvan - Centre Hospitalier Universitaire, Brest
  - Cabinet d'Oncologie - Hôpital Privé Sainte Marie, Chalon-sur-Saône
  - Centre Hospitalier de Cholet, Cholet
  - Hôpital Privé Drôme Ardèche - Clinique Pasteur, Guilherand-Granges
  - Hôpital Louis Pasteur, Le Coudray
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier Universitaire Dupuytren, Limoges
  - CHU Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - institut Paoli Calmette, Marseille
  - Centre Azuréen de Cancérologie, Mougins
  - Centre d'oncologie de Gentilly, Nancy
  - Centre Hospitalier Régional, Orléans
  - Hôpital Tenon, Paris
  - Hôpital de la Milétrie - Centre Hospitalier Universitaire de Poitiers - Pôle Régional de Cancérologie, Poitiers
  - Clinique Courlancy, Reims
  - Institut Jean Godinot, Reims
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - Clinique de l'Alliance, Saint-Cyr-sur-Loire
  - ICO Centre René Gauducheau, Saint-Herblain
  - Clinique de l'Union, Saint-Jean
  - GHPSO - Site Senlis, Senlis
  - Centre de Radiothérapie - Clinique Sainte-Anne, Strasbourg
  - Clinique Saint Jean, Toulon
  - Institut Claudius Regaud, Toulouse
  - Institut de Cancérologie Gustave Roussy, Villejuif

REFERENCES:
- [Result] Selle F, Heudel PE, Hardy-Bessard AC, Pozet A, Meunier J, Gladieff L, Lotz JP, Provansal M, Augereau P, Berton D, Bonichon-Lamichhane N, Orfeuvre H, Pautier P, Kalbacher E, Tazi Y, Spaeth D. GINECO Prospective Non-interventional PROSPECTYON Study: Trabectedin Plus Pegylated Liposomal Doxorubicin for Platinum-sensitive Recurrent Ovarian Cancer. Anticancer Res. 2020 Jul;40(7):3939-3945. doi: 10.21873/anticanres.14385. PMID 32620635